CLINICAL TRIAL: NCT03774940
Title: Neutrophil and Lymphocyte Counts and the Neutrophil-to-lymphocyte Ratio as a Predictor of Fever Following Percutaneous Nephrolithotomy in Patients Without Risk Factors
Brief Title: Blood Parameters as a Predictor of Fever After Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Assoc.Prof., TC Erciyes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013/198
Record Dates: First submitted 2018-12-09; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Urinary Tract Infection Bacterial; Nephrolithiasis
Keywords: fever; bacteremia; lymphocytes; percutaneous nephrolithotomy; neutrophil-lymphocyte ratio
MeSH Terms: conditions — Nephrolithiasis; Fever; Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fever (Experimental): patients that have fever after PNL
  Interventions: Diagnostic Test: peripheric blood count
- No fever (Active Comparator): Patients without fever after PNL
  Interventions: Diagnostic Test: peripheric blood count

INTERVENTIONS:
Diagnostic Test: peripheric blood count — preoperative peripheric blood count

SUMMARY:
To investigate the relationship between neutrophil count, lymphocyte count, neutrophil-to-lymphocyte count ratio (NLR), and postoperative fever in patients undergoing percutaneous nephrolithotomy (PNL).

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PNL) is a minimally invasive treatment commonly used for renal calculi. However, the prevalence of postoperative fever is reported to be 16.7%-35%, even with appropriate prophylactic antibiotic therapy and a sterile urine culture. The most probable causes are urinary extravasation and bacteremia. Although it is important to postoperatively isolate the causative bacteria, bacterial isolation may not always be possible, and urinary and blood cultures may prove negative. In addition, establishing the etiology of fever could be time-consuming and the techniques involved may generate pseudo-negative results owing to several factors, especially the antibiotics used prophylactically. This can result in a prolonged hospital stay and increased the cost of patient care.

The most commonly used parameters for the early diagnosis of bacterial infections, despite their limited use, are C-reactive protein, white blood cell count, and neutrophil count . Superior parameters include procalcitonin, pro-adrenomedullin, interleukin (IL)-6, and IL-8, but their use is limited by their lack of availability in some centers and their higher costs. Recently, the ratio of neutrophil count to lymphocyte count (NLR) has been proposed as an effective, simple, and useful biomarker for the early diagnosis of bacterial infections. However, these tests are used after the emergence of fever. As yet, no single parameter has been proposed for predicting postoperative fever in the absence of preoperative factors known to cause fever.

The aim of this study was to investigate whether neutrophil count, lymphocyte count, and NLR obtained from routine preoperative blood tests could be used in predicting fever following PNL in patients with no risk factors for infection.

ELIGIBILITY:
Inclusion Criteria:

* underwent PNL operation
* preoperative white blood cell count between 4,000 and 12,000/µL

Exclusion Criteria:

* preoperative urinary system obstruction
* proliferation in preoperative and/or postoperative urine culture
* preoperative and/or postoperative blood transfusions
* a preoperative urinary diversion and/or intervention
* the presence of a postoperative residual stone
* the presence of malignancy,
* the presence of a hematologic disease.
* patients with postoperative complications graded as Clavien 2 and above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
White blood cell count | preoperative
  white blood cell count
Neutrophil count | preoperative
  neutrophil count
N/L | preoperative
  ratio of neutrophil count to lymphocyte count
Lymphocyte count | preoperative
  Lymphocyte count

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Demirtas, MD, Principal Investigator — Erciyes University Faculty of Medicine
Locations (1):
- Erciyes University Faculty of Medicine Department of Urology, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Draga RO, Kok ET, Sorel MR, Bosch RJ, Lock TM. Percutaneous nephrolithotomy: factors associated with fever after the first postoperative day and systemic inflammatory response syndrome. J Endourol. 2009 Jun;23(6):921-7. doi: 10.1089/end.2009.0041. PMID 19473071
- [Background] Cadeddu JA, Chen R, Bishoff J, Micali S, Kumar A, Moore RG, Kavoussi LR. Clinical significance of fever after percutaneous nephrolithotomy. Urology. 1998 Jul;52(1):48-50. doi: 10.1016/s0090-4295(98)00146-0. PMID 9671869
- [Background] Sharifi Aghdas F, Akhavizadegan H, Aryanpoor A, Inanloo H, Karbakhsh M. Fever after percutaneous nephrolithotomy: contributing factors. Surg Infect (Larchmt). 2006 Aug;7(4):367-71. doi: 10.1089/sur.2006.7.367. PMID 16978080
- [Background] Nuutila J, Lilius EM. Distinction between bacterial and viral infections. Curr Opin Infect Dis. 2007 Jun;20(3):304-10. doi: 10.1097/QCO.0b013e3280964db4. PMID 17471042
- [Background] Lutfiyya MN, Henley E, Chang LF, Reyburn SW. Diagnosis and treatment of community-acquired pneumonia. Am Fam Physician. 2006 Feb 1;73(3):442-50. PMID 16477891
- [Background] Shapiro MF, Greenfield S. The complete blood count and leukocyte differential count. An approach to their rational application. Ann Intern Med. 1987 Jan;106(1):65-74. doi: 10.7326/0003-4819-106-1-65. PMID 3538968
- [Background] Seebach JD, Morant R, Ruegg R, Seifert B, Fehr J. The diagnostic value of the neutrophil left shift in predicting inflammatory and infectious disease. Am J Clin Pathol. 1997 May;107(5):582-91. doi: 10.1093/ajcp/107.5.582. PMID 9128272
- [Background] Wyllie DH, Bowler IC, Peto TE. Bacteraemia prediction in emergency medical admissions: role of C reactive protein. J Clin Pathol. 2005 Apr;58(4):352-6. doi: 10.1136/jcp.2004.022293. PMID 15790696
- [Background] Chalupa P, Beran O, Herwald H, Kasprikova N, Holub M. Evaluation of potential biomarkers for the discrimination of bacterial and viral infections. Infection. 2011 Oct;39(5):411-7. doi: 10.1007/s15010-011-0126-4. Epub 2011 Jul 1. PMID 21720792
- [Background] de Jager CP, van Wijk PT, Mathoera RB, de Jongh-Leuvenink J, van der Poll T, Wever PC. Lymphocytopenia and neutrophil-lymphocyte count ratio predict bacteremia better than conventional infection markers in an emergency care unit. Crit Care. 2010;14(5):R192. doi: 10.1186/cc9309. Epub 2010 Oct 29. PMID 21034463
- [Background] Terradas R, Grau S, Blanch J, Riu M, Saballs P, Castells X, Horcajada JP, Knobel H. Eosinophil count and neutrophil-lymphocyte count ratio as prognostic markers in patients with bacteremia: a retrospective cohort study. PLoS One. 2012;7(8):e42860. doi: 10.1371/journal.pone.0042860. Epub 2012 Aug 9. PMID 22912753
- [Background] Mariappan P, Smith G, Moussa SA, Tolley DA. One week of ciprofloxacin before percutaneous nephrolithotomy significantly reduces upper tract infection and urosepsis: a prospective controlled study. BJU Int. 2006 Nov;98(5):1075-9. doi: 10.1111/j.1464-410X.2006.06450.x. PMID 17034608
- [Background] Dogan HS, Sahin A, Cetinkaya Y, Akdogan B, Ozden E, Kendi S. Antibiotic prophylaxis in percutaneous nephrolithotomy: prospective study in 81 patients. J Endourol. 2002 Nov;16(9):649-53. doi: 10.1089/089277902761402989. PMID 12490017
- [Background] Seyrek M, Binbay M, Yuruk E, Akman T, Aslan R, Yazici O, Berberoglu Y, Muslumanoglu AY. Perioperative prophylaxis for percutaneous nephrolithotomy: randomized study concerning the drug and dosage. J Endourol. 2012 Nov;26(11):1431-6. doi: 10.1089/end.2012.0242. Epub 2012 Aug 2. PMID 22612061
- [Background] Demirtas A, Yildirim YE, Sofikerim M, Kaya EG, Akinsal EC, Tombul ST, Ekmekcioglu O, Gulmez I. Comparison of infection and urosepsis rates of ciprofloxacin and ceftriaxone prophylaxis before percutaneous nephrolithotomy: a prospective and randomised study. ScientificWorldJournal. 2012;2012:916381. doi: 10.1100/2012/916381. Epub 2012 Dec 17. PMID 23319889
- [Background] Zahorec R. Ratio of neutrophil to lymphocyte counts--rapid and simple parameter of systemic inflammation and stress in critically ill. Bratisl Lek Listy. 2001;102(1):5-14. English, Slovak. PMID 11723675
- [Background] Goodman DA, Goodman CB, Monk JS. Use of the neutrophil:lymphocyte ratio in the diagnosis of appendicitis. Am Surg. 1995 Mar;61(3):257-9. PMID 7887542
- [Background] de Jager CP, Wever PC, Gemen EF, Kusters R, van Gageldonk-Lafeber AB, van der Poll T, Laheij RJ. The neutrophil-lymphocyte count ratio in patients with community-acquired pneumonia. PLoS One. 2012;7(10):e46561. doi: 10.1371/journal.pone.0046561. Epub 2012 Oct 1. PMID 23049706
- [Background] Tang K, Liu H, Jiang K, Ye T, Yan L, Liu P, Xia D, Chen Z, Xu H, Ye Z. Predictive value of preoperative inflammatory response biomarkers for metabolic syndrome and post-PCNL systemic inflammatory response syndrome in patients with nephrolithiasis. Oncotarget. 2017 Aug 18;8(49):85612-85627. doi: 10.18632/oncotarget.20344. eCollection 2017 Oct 17. PMID 29156745
- [Background] Cetinkaya M, Buldu I, Kurt O, Inan R. Platelet-to-Lymphocyte Ratio: A New Factor for Predicting Systemic Inflammatory Response Syndrome after Percutaneous Nephrolithotomy. Urol J. 2017 Aug 29;14(5):4089-4093. PMID 28853103
- [Background] Sen V, Bozkurt IH, Aydogdu O, Yonguc T, Yarimoglu S, Sen P, Koras O, Degirmenci T. Significance of preoperative neutrophil-lymphocyte count ratio on predicting postoperative sepsis after percutaneous nephrolithotomy. Kaohsiung J Med Sci. 2016 Oct;32(10):507-513. doi: 10.1016/j.kjms.2016.08.008. Epub 2016 Sep 9. PMID 27742034